CLINICAL TRIAL: NCT04630002
Title: Open-Label, Single-Sequence Study to Evaluate the Effects of Darunavir/Ritonavir and/or Etravirine on the Pharmacokinetics of GSK3640254 and the Effects of GSK3640254 on the Pharmacokinetics of Darunavir/Ritonavir and/or Etravirine in Heathy Adults
Brief Title: Drug-drug Interaction (DDI) Study of GSK3640254 With Darunavir/Ritonavir (DRV/RTV) and Etravirine (ETR)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 213054
Record Dates: First submitted 2020-11-11; First posted 2020-11-16 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: HIV Infections
Keywords: Darunavir; Ritonavir; Etravirine; GSK3640254; Pharmacokinetics
MeSH Terms: conditions — HIV Infections | interventions — GSK3640254; Darunavir; Ritonavir; etravirine

STUDY DESIGN:
Intervention Model Description: This is an open-label, single-sequence, multiple-dose and 3-cohort study.
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: GSK3640254 then DRV/RTV then GSK3640254 + DRV/RTV (Experimental): Cohort 1 will include 3 periods. In Period 1 GSK3640254 will be administered (Treatment A). In Period 2 DRV/RTV will be administered (Treatment B). In Period 3 GSK3640254 (Treatment A) and DRV/RTV (Treatment B) will be administered.
  Interventions: Drug: GSK3640254; Drug: Darunavir/Ritonavir (DRV/RTV)
- Cohort 2: GSK3640254 then ETR then GSK3640254 + ETR (Experimental): Cohort 2 will include 3 periods. In Period 1 GSK3640254 will be given (Treatment A). In Period 2 ETR will be given (Treatment C). In Period 3 GSK3640254 (Treatment A) and ETR (Treatment C) will be administered.
  Interventions: Drug: GSK3640254; Drug: Etravirine (ETR)
- Cohort 3: GSK3640254 then GSK3640254 + DRV/RTV + ETR (Experimental): Cohort 3 will include 2 periods. In Period 1 GSK3640254 will be administered (Treatment A). In Period 2 GSK3640254 (Treatment A), DRV/RTV (Treatment B), and ETR (Treatment C) will be administered.
  Interventions: Drug: GSK3640254; Drug: Darunavir/Ritonavir (DRV/RTV); Drug: Etravirine (ETR)

INTERVENTIONS:
Drug: GSK3640254 — GSK3640254 will be available as oral tablets.
Drug: Darunavir/Ritonavir (DRV/RTV) — DRV/RTV will be available as oral tablets.
  Arms: Cohort 1: GSK3640254 then DRV/RTV then GSK3640254 + DRV/RTV; Cohort 3: GSK3640254 then GSK3640254 + DRV/RTV + ETR
Drug: Etravirine (ETR) — ETR will be available as oral tablets.
  Arms: Cohort 2: GSK3640254 then ETR then GSK3640254 + ETR; Cohort 3: GSK3640254 then GSK3640254 + DRV/RTV + ETR

SUMMARY:
This is an open-label, single-sequence, multiple-dose, 3 cohort study to investigate the effects of DRV/RTV and/or ETR on the pharmacokinetics (PK) of GSK3640254 and the effects of GSK3640254 on the PK of DRV/RTV and/or ETR. This study will aid in understanding these interactions and resulting changes in exposure (if any) when given in combination with GSK3640254.

ELIGIBILITY:
Inclusion criteria:

* Participant must be 18 to 50 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring (history and screening ECG).
* Body weight more than or equal to (>=)50.0 kilograms (kg) (110 pounds [lbs]) for men and >=45.0 kg (99 lbs) for women and body mass index within the range 18.5 to 31.0 kilograms per square meter (kg/m^2) (inclusive).
* Male or female participants:

  1. Male participants should not engage in intercourse while confined in the study site. There is no need for an extended period of double barrier use or prolonged abstinence after study discharge.
  2. Female participants:

  (i) A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: Is not a woman of childbearing potential (WOCBP) OR Is a WOCBP and using a non-hormonal contraceptive method that is highly effective, with a failure rate of less than (<)1 percent (%) for 28 days before intervention, during the intervention period, and for at least 28 days after the last dose of study intervention. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.

(ii) A WOCBP must have a negative highly sensitive serum or urine pregnancy test at screening and check-in (Day -1).

* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the Informed consent form (ICF) and in this protocol.

Exclusion criteria:

* Participants with current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A pre-existing condition interfering with normal Gastrointestinal (GI) anatomy or motility (for example [e.g.], gastroesophageal reflux disease, gastric ulcers, gastritis) or hepatic and/or renal function that could interfere with the absorption, metabolism, and/or excretion of the study intervention or render the participant unable to take oral study intervention.
* Prior cholecystectomy surgery (prior appendectomy is acceptable).
* Clinically significant illness, including viral syndromes within 3 weeks of dosing.
* A participant with known or suspected active Coronavirus Disease-2019 (COVID-19) infection or contact with an individual with known COVID-19, within 14 days of study enrollment (World Health Organization [WHO] definitions).
* Any history of significant underlying psychiatric disorder, including, but not limited to, schizophrenia, bipolar disorder with or without psychotic symptoms, other psychotic disorders, or schizotypal (personality) disorder.
* Any history of major depressive disorder with or without suicidal features, or anxiety disorders that required medical intervention (pharmacologic or not) such as hospitalization or other inpatient treatment and/or chronic (more than [>]6 months) outpatient treatment. Participants with other conditions such as adjustment disorder or dysthymia that have required shorter term medical therapy (<6 months) without inpatient treatment and are currently well-controlled clinically or resolved may be considered for entry after discussion and agreement with the ViiV Healthcare/GlaxoSmithKline (VH/GSK) medical monitor.
* Any pre-existing physical or other psychiatric condition (including alcohol or drug abuse), which, in the opinion of the investigator (with or without psychiatric evaluation), could interfere with the participant's ability to comply with the dosing schedule and protocol evaluations or which might compromise the safety of the participant.
* Medical history of cardiac arrhythmias, prior myocardial infarction in the past 3 months, or cardiac disease or a family or personal history of long QT syndrome.
* Presence of hepatitis B surface antigen at screening or within 3 months prior to starting study intervention.
* Positive hepatitis C antibody test result at screening or within 3 months prior to starting study intervention.
* Positive Human immunodeficiency virus (HIV)-1 and -2 antigen/antibody immunoassay at screening.
* Alanine aminotransferase (ALT) >1.5 times upper limit of normal (ULN). A single repeat of ALT is allowed within a single screening period to determine eligibility.
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat of any laboratory abnormality is allowed within a single screening period to determine eligibility.
* Any acute laboratory abnormality at screening which, in the opinion of the investigator, should preclude participation in the study of an investigational compound.
* Any Grade 2 to 4 laboratory abnormality at screening, with the exception of creatine phosphokinase (CPK), lipid abnormalities (e.g., total cholesterol, triglycerides), and ALT (described above), will exclude a participant from the study unless the investigator can provide a compelling explanation for the laboratory result(s) and has the assent of the sponsor. A single repeat of any laboratory abnormality is allowed within a single screening period to determine eligibility.
* Urine drug screen positive (showing presence of): amphetamines, barbiturates, cannabinoids, cocaine, or phencyclidine, or non-prescribed opiates, oxycodone, benzodiazepines, methadone, Methylenedioxymethamphetamine (MDMA), methamphetamines, or tricyclic antidepressants at screening or before the first dose of study intervention.
* Unable to refrain from the use of prescription or nonprescription drugs including vitamins, herbal and dietary supplements (including Saint [St] John's wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study intervention and for the duration of the study.
* Treatment with any vaccine within 30 days prior to receiving study intervention.
* Unwillingness to abstain from excessive consumption of any food or drink containing grapefruit and grapefruit juice, Seville oranges, blood oranges, or pomelos or their fruit juices within 7 days prior to the first dose of study intervention(s) until the end of the study.
* Participation in another concurrent clinical study or prior clinical study (with the exception of imaging trials) prior to the first dosing day in the current study: 30 days, 5 half-lives, or twice the duration of the biological effect of the study intervention (whichever is longer).
* Prior exposure to GSK3640254 or prior intolerance to DRV/RTV or ETR in this or another clinical study.
* Prior intolerance to any other study medications: DRV/RTV or ETR.
* Where participation in the study would result in donation of blood or blood products in excess of 500 milliliters (mL) within 56 days.
* Any positive (abnormal) response confirmed by the investigator on a screening clinician- or qualified designee-administered Columbia-Suicide Severity Rating Scale (C-SSRS).
* Systolic blood pressure <100 millimeters of mercury (mm Hg). Up to 2 repeats are allowed for confirmation.
* Any significant arrhythmia or ECG finding (e.g., prior myocardial infarction in the past 3 months, symptomatic bradycardia, non-sustained or sustained atrial arrhythmias, non-sustained or sustained ventricular tachycardia, any degree of atrioventricular block, or conduction abnormality) which, in the opinion of the investigator or VH/GSK medical monitor, will interfere with the safety for the individual participant.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination):

  1. Heart rate: <50 or >100 beats per minute (bpm).
  2. PR interval >200 milliseconds (ms).
  3. Corrected QT interval (QTc) >450 ms.
* History of regular alcohol consumption within 6 months of the study, defined as an average weekly intake of >14 units. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine, or 1 (25 mL) measure of spirits.
* Unable to refrain from tobacco or nicotine-containing products within 3 months prior to screening.
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2021-10-02 (Actual); Study Completion 2021-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
ViiV will assess requests from qualified researchers for anonymized individual patient-level data (IPD) and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf

REFERENCES:
- [Background] Zhang Y, Joshi S, Yazdani P, Zhan J, Wen B, Bainbridge V, Ballesteros-Perez A, Gartland M, Lataillade M. Pharmacokinetics and tolerability of the maturation inhibitor GSK3640254 coadministered with darunavir/ritonavir and/or etravirine in healthy adults. Br J Clin Pharmacol. 2024 Jan;90(1):274-285. doi: 10.1111/bcp.15893. Epub 2023 Sep 20. PMID 37621050

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in the United States.
Pre-assignment Details: A total of 54 participants (19 in Cohort 1, 19 in Cohort 2 and 16 in Cohort 3) were enrolled in the study (Safety Population: It comprised of all participants who received at least 1 dose of study medication).
Groups:
- Cohort 1: GSK3640254 Then DRV/RTV Then GSK3640254 + DRV/RTV: Participants received GSK3640254 200 milligram (mg) tablets once daily on Days 1 to 7 in treatment period 1 followed by Darunavir/Ritonavir (DRV/RTV) 600/100 mg tablets twice daily on Days 12 to 21 in treatment period 2. There was a washout period on Days 8 to 11 between treatment periods 1 and 2. Participants also received GSK3640254 200 mg tablets once daily along with DRV/RTV 600/100 mg tablets twice daily on Days 22 to 31 in treatment period 3.
- Cohort 2: GSK3640254 Then ETR Then GSK3640254 + ETR: Participants received GSK3640254 200 mg tablets once daily on Days 1 to 7 in treatment period 1 followed by Etravirine (ETR) 200 mg tablets twice daily on Days 12 to 21 in treatment period 2. There was a washout period on Days 8 to 11 between treatment periods 1 and 2. Participants also received GSK3640254 200 mg tablets once daily along with ETR 200 mg tablets twice daily on Days 22 to 31 in treatment period 3.
- Cohort 3: GSK3640254 Then GSK3640254 + DRV/RTV + ETR: Participants received GSK3640254 200 mg tablets once daily on Days 1 to 7 in treatment period 1. Participants received GSK3640254 200 mg tablets once daily along with DRV/RTV 600/100 mg tablets twice daily and ETR 200 mg tablets twice daily on Days 8 to 21 in treatment period 2.
Period: Cohort 1:Treatment Period 1(Days 1 to 7)
Arm/Group | Cohort 1: GSK3640254 Then DRV/RTV Then GSK3640254 + DRV/RTV | Cohort 2: GSK3640254 Then ETR Then GSK3640254 + ETR | Cohort 3: GSK3640254 Then GSK3640254 + DRV/RTV + ETR
Started | 19 | 0 | 0
Completed | 19 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Cohort 1:Washout Period (Days 8 to 11)
Arm/Group | Cohort 1: GSK3640254 Then DRV/RTV Then GSK3640254 + DRV/RTV | Cohort 2: GSK3640254 Then ETR Then GSK3640254 + ETR | Cohort 3: GSK3640254 Then GSK3640254 + DRV/RTV + ETR
Started | 19 | 0 | 0
Completed | 19 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Cohort1:Treatment Period2(Days 12 to 21)
Arm/Group | Cohort 1: GSK3640254 Then DRV/RTV Then GSK3640254 + DRV/RTV | Cohort 2: GSK3640254 Then ETR Then GSK3640254 + ETR | Cohort 3: GSK3640254 Then GSK3640254 + DRV/RTV + ETR
Started | 19 | 0 | 0
Completed | 17 | 0 | 0
Not Completed | 2 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0
Period: Cohort1:Treatment Period3(Days 22 to 31)
Arm/Group | Cohort 1: GSK3640254 Then DRV/RTV Then GSK3640254 + DRV/RTV | Cohort 2: GSK3640254 Then ETR Then GSK3640254 + ETR | Cohort 3: GSK3640254 Then GSK3640254 + DRV/RTV + ETR
Started | 17 | 0 | 0
Completed | 15 | 0 | 0
Not Completed | 2 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Period: Cohort 2:Treatment Period 1(Days 1 to 7)
Arm/Group | Cohort 1: GSK3640254 Then DRV/RTV Then GSK3640254 + DRV/RTV | Cohort 2: GSK3640254 Then ETR Then GSK3640254 + ETR | Cohort 3: GSK3640254 Then GSK3640254 + DRV/RTV + ETR
Started | 0 | 19 | 0
Completed | 0 | 19 | 0
Not Completed | 0 | 0 | 0
Period: Cohort 2: Washout Period (Days 8 to 11)
Arm/Group | Cohort 1: GSK3640254 Then DRV/RTV Then GSK3640254 + DRV/RTV | Cohort 2: GSK3640254 Then ETR Then GSK3640254 + ETR | Cohort 3: GSK3640254 Then GSK3640254 + DRV/RTV + ETR
Started | 0 | 19 | 0
Completed | 0 | 19 | 0
Not Completed | 0 | 0 | 0
Period: Cohort2:Treatment Period2(Days 12 to 21)
Arm/Group | Cohort 1: GSK3640254 Then DRV/RTV Then GSK3640254 + DRV/RTV | Cohort 2: GSK3640254 Then ETR Then GSK3640254 + ETR | Cohort 3: GSK3640254 Then GSK3640254 + DRV/RTV + ETR
Started | 0 | 19 | 0
Completed | 0 | 17 | 0
Not Completed | 0 | 2 | 0
Not completed — Physician Decision | 0 | 2 | 0
Period: Cohort2:Treatment Period3(Days 22 to 31)
Arm/Group | Cohort 1: GSK3640254 Then DRV/RTV Then GSK3640254 + DRV/RTV | Cohort 2: GSK3640254 Then ETR Then GSK3640254 + ETR | Cohort 3: GSK3640254 Then GSK3640254 + DRV/RTV + ETR
Started | 0 | 17 | 0
Completed | 0 | 14 | 0
Not Completed | 0 | 3 | 0
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 0
Period: Cohort 3:Treatment Period 1(Days 1 to 7)
Arm/Group | Cohort 1: GSK3640254 Then DRV/RTV Then GSK3640254 + DRV/RTV | Cohort 2: GSK3640254 Then ETR Then GSK3640254 + ETR | Cohort 3: GSK3640254 Then GSK3640254 + DRV/RTV + ETR
Started | 0 | 0 | 16
Completed | 0 | 0 | 16
Not Completed | 0 | 0 | 0
Period: Cohort 3:Treatment Period2(Days 8 to 21)
Arm/Group | Cohort 1: GSK3640254 Then DRV/RTV Then GSK3640254 + DRV/RTV | Cohort 2: GSK3640254 Then ETR Then GSK3640254 + ETR | Cohort 3: GSK3640254 Then GSK3640254 + DRV/RTV + ETR
Started | 0 | 0 | 16
Completed | 0 | 0 | 14
Not Completed | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were reported for Safety Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: GSK3640254 Then DRV/RTV Then GSK3640254 + DRV/RTV | Cohort 2: GSK3640254 Then ETR Then GSK3640254 + ETR | Cohort 3: GSK3640254 Then GSK3640254 + DRV/RTV + ETR | Total
Number analyzed (Participants) | 19 | 19 | 16 | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.3 (5.98) | 31.2 (6.18) | 32.0 (9.21) | 32.5 (7.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 2 | 11
  Male | 14 | 15 | 14 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN-CENTRAL/SOUTH ASIAN HERITAGE (H) | 0 | 1 | 0 | 1
  ASIAN-JAPANESE H/EAST ASIAN H/SOUTH EAST ASIAN H | 0 | 1 | 0 | 1
  BLACK (BLA) OR AFRICAN AMERICAN (AFR AME) | 10 | 8 | 6 | 24
  WHITE-ARABIC NORTH AFR WHITE H | 1 | 2 | 1 | 4
  WHITE-CAUCASIAN EUROPEAN WHITE H | 7 | 7 | 9 | 23
  AME INDIAN OR ALASKA NATIVE &BLA OR AFR AMR &WHITE | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Area Under the Plasma Concentration-time Curve From Time Zero to the End of the Dosing Interval at Steady State (AUC[0-tau]) of GSK3640254
Description: Blood samples were collected at indicated time points. Pharmacokinetic analysis was conducted using standard non-compartmental methods.
Time Frame: Pre-dose and 0.5 Hours, 1 Hour, 1.5 Hours, 2 Hours, 3 Hours, 4 Hours, 6 Hours, 8 Hours, 12 Hours, 16 Hours, 24 Hours post-dose in Treatment Periods 1 and 3
Population: Pharmacokinetic Parameter Population comprised of all participants who underwent plasma pharmacokinetic sampling and had at least 1 evaluable Pharmacokinetic parameter estimated. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Groups:
- Cohort 1: GSK3640254 200 mg: Participants received GSK3640254 200 mg tablets once daily on Days 1 to 7 in Treatment Period 1 of Cohort 1 of the study.
- Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg: Participants received GSK3640254 200 mg tablets once daily along with DRV/RTV 600/100 mg tablets twice daily on Days 22 to 31 in Treatment Period 3 of Cohort 1 of the study.
Arm/Group | Cohort 1: GSK3640254 200 mg | Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg
Number analyzed (Participants) | 16 | 15
Hours*micrograms per milliliter | 27.03 (33.7) | 30.70 (33.6)
Statistical Analysis 1: Comparison: Cohort 1: GSK3640254 200 mg vs Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg; Test type: Other; Ratio of geometric least square means = 1.137, 90% CI 2-sided [0.9990 to 1.293] — A linear mixed-effects model with period as a fixed effect, participant as a random effect, and measurements within participant as repeated measures was performed on the log-transformed parameter AUC(0-tau)

2. Primary Outcome: Cohort 1: Maximum Observed Concentration (Cmax) of GSK3640254
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Cohort 1: GSK3640254 200 mg | Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg
Number analyzed (Participants) | 16 | 15
Micrograms per milliliter | 1.752 (39.1) | 1.863 (41.0)
Statistical Analysis 1: Comparison: Cohort 1: GSK3640254 200 mg vs Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg; Test type: Other; Ratio of geometric least square means = 1.068, 90% CI 2-sided [0.9185 to 1.242] — A linear mixed-effects model with period as a fixed effect, participant as a random effect, and measurements within participant as repeated measures was performed on the log-transformed parameter Cmax

3. Primary Outcome: Cohort 1: AUC(0-tau) of DRV
Description: as for outcome 1
Time Frame: Pre-dose and 0.5 Hours, 1 Hour, 1.5 Hours, 2 Hours, 3 Hours, 4 Hours, 6 Hours, 8 Hours, 12 Hours post-dose in Treatment Periods 2 and 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Groups:
- Cohort 1: DRV/RTV 600/100 mg: Participants received DRV/RTV 600/100 mg tablets twice daily on Days 12 to 21 in Treatment Period 2 of Cohort 1 of the study.
- Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg: Participants received GSK3640254 200 mg tablets once daily plus DRV/RTV 600/100 mg tablets twice daily on Days 22 to 31 in Treatment Period 3 of Cohort 1 of the study.
Arm/Group | Cohort 1: DRV/RTV 600/100 mg | Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg
Number analyzed (Participants) | 16 | 15
Hours*micrograms per milliliter | 57.47 (25.7) | 53.37 (22.1)
Statistical Analysis 1: Comparison: Cohort 1: DRV/RTV 600/100 mg vs Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg; Test type: Other; Ratio of geometric least square means = 0.9891, 90% CI 2-sided [0.9313 to 1.051] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Cohort 1: Cmax of DRV
Description: as for outcome 1
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Cohort 1: DRV/RTV 600/100 mg | Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg
Number analyzed (Participants) | 16 | 15
Micrograms per milliliter | 7.037 (24.4) | 7.268 (21.7)
Statistical Analysis 1: Comparison: Cohort 1: DRV/RTV 600/100 mg vs Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg; Test type: Other; Ratio of geometric least square means = 1.050, 90% CI 2-sided [0.9816 to 1.122] — [estimate comment as in outcome 2, analysis 1]

5. Primary Outcome: Cohort 1: AUC(0-tau) of RTV
Description: as for outcome 1
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours* micrograms per milliliter
Arm/Group | Cohort 1: DRV/RTV 600/100 mg | Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg
Number analyzed (Participants) | 16 | 15
Hours* micrograms per milliliter | 7.303 (48.7) | 7.790 (45.9)
Statistical Analysis 1: Comparison: Cohort 1: DRV/RTV 600/100 mg vs Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg; Test type: Other; Ratio of geometric least square means = 1.102, 90% CI 2-sided [1.025 to 1.185] — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: Cohort 1: Cmax of RTV
Description: as for outcome 1
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Cohort 1: DRV/RTV 600/100 mg | Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg
Number analyzed (Participants) | 16 | 15
Micrograms per milliliter | 1.178 (43.1) | 1.306 (36.6)
Statistical Analysis 1: Comparison: Cohort 1: DRV/RTV 600/100 mg vs Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg; Test type: Other; Ratio of geometric least square means = 1.120, 90% CI 2-sided [0.9947 to 1.260] — [estimate comment as in outcome 2, analysis 1]

7. Primary Outcome: Cohort 2: AUC(0-tau) of GSK3640254
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Groups:
- Cohort 2: GSK3640254 200 mg: Participants received GSK3640254 200 mg tablets once daily on Days 1 to 7 in Treatment period 1 of Cohort 2 of the study.
- Cohort 2: GSK3640254 200 mg + ETR 200 mg: Participants received GSK3640254 200 mg tablets once daily along with ETR 200 mg tablets twice daily on Days 22 to 31 in Treatment Period 3 of Cohort 2 of the study.
Arm/Group | Cohort 2: GSK3640254 200 mg | Cohort 2: GSK3640254 200 mg + ETR 200 mg
Number analyzed (Participants) | 16 | 15
Hours*micrograms per milliliter | 27.86 (27.8) | 14.73 (26.5)
Statistical Analysis 1: Comparison: Cohort 2: GSK3640254 200 mg vs Cohort 2: GSK3640254 200 mg + ETR 200 mg; Test type: Other; Ratio of geometric least square means = 0.5299, 90% CI 2-sided [0.4801 to 0.5848] — [estimate comment as in outcome 1, analysis 1]

8. Primary Outcome: Cohort 2: Cmax of GSK3640254
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Cohort 2: GSK3640254 200 mg | Cohort 2: GSK3640254 200 mg + ETR 200 mg
Number analyzed (Participants) | 16 | 15
Micrograms per milliliter | 1.889 (38.2) | 1.136 (28.5)
Statistical Analysis 1: Comparison: Cohort 2: GSK3640254 200 mg vs Cohort 2: GSK3640254 200 mg + ETR 200 mg; Test type: Other; Ratio of geometric least square means = 0.6001, 90% CI 2-sided [0.5271 to 0.6833] — [estimate comment as in outcome 2, analysis 1]

9. Primary Outcome: Cohort 2: AUC(0-tau) of ETR
Description: as for outcome 1
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Groups:
- Cohort 2: ETR 200 mg: Participants received ETR 200 mg tablets twice daily on Days 12 to 21 Treatment Period 2 of Cohort 2 of the study.
Arm/Group | Cohort 2: ETR 200 mg | Cohort 2: GSK3640254 200 mg + ETR 200 mg
Number analyzed (Participants) | 16 | 15
Hours*micrograms per milliliter | 8.340 (36.0) | 9.791 (32.8)
Statistical Analysis 1: Comparison: Cohort 2: ETR 200 mg vs Cohort 2: GSK3640254 200 mg + ETR 200 mg; Test type: Other; Ratio of geometric least square means = 1.144, 90% CI 2-sided [1.082 to 1.210] — [estimate comment as in outcome 1, analysis 1]

10. Primary Outcome: Cohort 2: Cmax of ETR
Description: as for outcome 1
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Cohort 2: ETR 200 mg | Cohort 2: GSK3640254 200 mg + ETR 200 mg
Number analyzed (Participants) | 16 | 15
Micrograms per milliliter | 0.9749 (35.1) | 1.102 (33.0)
Statistical Analysis 1: Comparison: Cohort 2: ETR 200 mg vs Cohort 2: GSK3640254 200 mg + ETR 200 mg; Test type: Other; Ratio of geometric least square means = 1.104, 90% CI 2-sided [1.026 to 1.187] — [estimate comment as in outcome 2, analysis 1]

11. Primary Outcome: Cohort 3: AUC(0-tau) of GSK3640254
Description: as for outcome 1
Time Frame: Pre-dose and 0.5 Hours, 1 Hour, 1.5 Hours, 2 Hours, 3 Hours, 4 Hours, 6 Hours, 8 Hours, 12 Hours, 16 Hours, 24 Hours post-dose in Treatment Periods 1 and 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Groups:
- Cohort 3: GSK3640254 200 mg: Participants received GSK3640254 200 mg tablets once daily on Days 1 to 7 in Treatment Period 1 of Cohort 3 of the study.
- Cohort 3: GSK3640254 200 mg+ DRV/RTV 600/100 mg+ ETR 200 mg: Participants received GSK3640254 200 mg tablets once daily along with DRV/RTV 600/100 mg tablets twice daily and ETR 200 mg tablets twice daily on Days 8 to 21 in Treatment Period 2 of Cohort 3 of the study.
Arm/Group | Cohort 3: GSK3640254 200 mg | Cohort 3: GSK3640254 200 mg+ DRV/RTV 600/100 mg+ ETR 200 mg
Number analyzed (Participants) | 16 | 14
Hours*micrograms per milliliter | 24.99 (34.7) | 22.78 (34.3)
Statistical Analysis 1: Comparison: Cohort 3: GSK3640254 200 mg vs Cohort 3: GSK3640254 200 mg+ DRV/RTV 600/100 mg+ ETR 200 mg; Test type: Other; Ratio of geometric least square means = 0.9435, 90% CI 2-sided [0.8147 to 1.093] — [estimate comment as in outcome 1, analysis 1]

12. Primary Outcome: Cohort 3: Cmax of GSK3640254
Description: as for outcome 1
Time Frame: as for outcome 11
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Cohort 3: GSK3640254 200 mg | Cohort 3: GSK3640254 200 mg+ DRV/RTV 600/100 mg+ ETR 200 mg
Number analyzed (Participants) | 16 | 14
Micrograms per milliliter | 1.578 (34.8) | 1.383 (32.5)
Statistical Analysis 1: Comparison: Cohort 3: GSK3640254 200 mg vs Cohort 3: GSK3640254 200 mg+ DRV/RTV 600/100 mg+ ETR 200 mg; Test type: Other; Ratio of geometric least square means = 0.8928, 90% CI 2-sided [0.7467 to 1.068] — [estimate comment as in outcome 2, analysis 1]

13. Secondary Outcome: Cohort 1: Plasma Concentration at the End of the Dosing Interval (Ctau) of DRV
Description: as for outcome 1
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Cohort 1: DRV/RTV 600/100 mg | Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg
Number analyzed (Participants) | 16 | 15
Micrograms per milliliter | 2.957 (37.0) | 2.637 (36.5)

14. Secondary Outcome: Cohort 1: Time of Maximum Observed Concentration (Tmax) of DRV
Description: as for outcome 1
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Groups:
- Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg: Participants received GSK3640254 200 mg tablets once daily along with DRV/RTV 600/100 mg tablets twice daily on Days 22 to 31 in Treatment Period 3 of Cohort 1 of the
Arm/Group | Cohort 1: DRV/RTV 600/100 mg | Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg
Number analyzed (Participants) | 16 | 15
Hours | 3.000 [1.50 to 4.00] | 3.000 [1.57 to 4.00]

15. Secondary Outcome: Cohort 1: Ctau of RTV
Description: as for outcome 1
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Cohort 1: DRV/RTV 600/100 mg | Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg
Number analyzed (Participants) | 16 | 15
Micrograms per milliliter | 0.3194 (77.4) | 0.3314 (91.1)

16. Secondary Outcome: Cohort 1: Tmax of RTV
Description: as for outcome 1
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: DRV/RTV 600/100 mg | Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg
Number analyzed (Participants) | 16 | 15
Hours | 4.000 [2.00 to 6.00] | 4.000 [2.00 to 4.00]

17. Secondary Outcome: Cohort 1: Ctau of GSK3640254
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Cohort 1: GSK3640254 200 mg | Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg
Number analyzed (Participants) | 16 | 15
Micrograms per milliliter | 0.8152 (34.5) | 0.9530 (35.2)

18. Secondary Outcome: Cohort 1: Tmax of GSK3640254
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: GSK3640254 200 mg | Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg
Number analyzed (Participants) | 16 | 15
Hours | 4.000 [1.50 to 8.00] | 4.000 [1.50 to 11.93]

19. Secondary Outcome: Cohort 2: Ctau of ETR
Description: as for outcome 1
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Cohort 2: ETR 200 mg | Cohort 2: GSK3640254 200 mg + ETR 200 mg
Number analyzed (Participants) | 16 | 15
Micrograms per milliliter | 0.4705 (37.8) | 0.5837 (33.1)

20. Secondary Outcome: Cohort 2: Tmax of ETR
Description: as for outcome 1
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 2: ETR 200 mg | Cohort 2: GSK3640254 200 mg + ETR 200 mg
Number analyzed (Participants) | 16 | 15
Hours | 3.500 [2.00 to 6.00] | 4.000 [2.00 to 8.00]

21. Secondary Outcome: Cohort 2: Ctau of GSK3640254
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Cohort 2: GSK3640254 200 mg | Cohort 2: GSK3640254 200 mg + ETR 200 mg
Number analyzed (Participants) | 16 | 15
Micrograms per milliliter | 0.7706 (36.3) | 0.3901 (50.2)

22. Secondary Outcome: Cohort 2: Tmax of GSK3640254
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 2: GSK3640254 200 mg | Cohort 2: GSK3640254 200 mg + ETR 200 mg
Number analyzed (Participants) | 16 | 15
Hours | 4.000 [2.00 to 8.00] | 3.000 [2.00 to 6.00]

23. Secondary Outcome: Cohort 1: Number of Participants With Serious Adverse Events (SAEs) and Non-serious Adverse Events (Non-SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or other situations as per medical or scientific judgment. Adverse events which were not Serious were considered as Non-Serious adverse events.
Time Frame: Up to Day 35
Population: Safety Population comprised of all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: GSK3640254 200 mg | Cohort 1: DRV/RTV 600/100 mg | Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg
Number analyzed (Participants) | 19 | 16 | 15
Participants
  SAE | 0 | 0 | 0
  non-SAE | 6 | 4 | 5

24. Secondary Outcome: Cohort 2: Number of Participants With SAEs and Non-SAEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or other situations as per medical or scientific judgment. Adverse events which were not Serious were considered as Non-Serious adverse events.
Time Frame: Up to Day 36
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: GSK3640254 200 mg | Cohort 2: ETR 200 mg | Cohort 2: GSK3640254 200 mg + ETR 200 mg
Number analyzed (Participants) | 19 | 16 | 16
Participants
  SAE | 0 | 0 | 0
  non-SAE | 3 | 4 | 7

25. Secondary Outcome: Cohort 3: Number of Participants With SAEs and Non-SAEs
Description: as for outcome 24
Time Frame: Up to Day 26
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: GSK3640254 200 mg | Cohort 3: GSK3640254 200 mg+ DRV/RTV 600/100 mg+ ETR 200 mg
Number analyzed (Participants) | 16 | 15
Participants
  SAE | 0 | 0
  non-SAE | 1 | 8

26. Secondary Outcome: Cohort 1: Number of Participants With AEs Leading to Discontinuations and Deaths
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Number of participants with AEs leading to discontinuations and deaths were reported.
Time Frame: Up to Day 35
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: GSK3640254 200 mg | Cohort 1: DRV/RTV 600/100 mg | Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg
Number analyzed (Participants) | 19 | 16 | 15
Participants
  AEs leading to discontinuations | 0 | 1 | 0
  AES leading to deaths | 0 | 0 | 0

27. Secondary Outcome: Cohort 2: Number of Participants With AEs Leading to Discontinuations and Deaths
Description: as for outcome 26
Time Frame: Up to Day 36
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: GSK3640254 200 mg | Cohort 2: ETR 200 mg | Cohort 2: GSK3640254 200 mg + ETR 200 mg
Number analyzed (Participants) | 19 | 16 | 16
Participants
  AEs leading to discontinuations | 0 | 0 | 1
  AES leading to deaths | 0 | 0 | 0

28. Secondary Outcome: Cohort 3: Number of Participants With AEs Leading to Discontinuations and Deaths
Description: as for outcome 26
Time Frame: Up to Day 26
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: GSK3640254 200 mg | Cohort 3: GSK3640254 200 mg+ DRV/RTV 600/100 mg+ ETR 200 mg
Number analyzed (Participants) | 16 | 15
Participants
  AEs leading to discontinuations | 0 | 1
  AES leading to deaths | 0 | 0

29. Secondary Outcome: Cohort 1: Number of Participants With Grade Increase Post-Baseline Relative to Baseline in Hematology Parameters
Description: Blood samples were collected for analysis of hematology parameters. Laboratory abnormalities were graded according to Division of Acquired Immunodeficiency Syndrome (DAIDS) grading table Version 2.1. For Hemoglobin Low, Grade 3: 7.0 to <9.0 Grams per deciliter (g/dL) (males) and 6.5 to <8.5 g/dL (females),Grade 4: <7.0 g/dL (males) and <6.5 g/dL (females); Leukocytes Low, Grade 3: 1000 to 1499 cells per cubic millimeter (cells/mm^3),Grade 4: <1000 cells/mm^3; Lymphocytes Low, Grade 3: 350 to <500 cells per liter (cells/L),Grade 4: <350 cells/L; Neutrophils Low, Grade 3: 400 to 599 cells/mm^3, Grade 4: <400 cells/mm^3; Platelets Low, Grade 3: 25,000 to <50,000 cells/mm^3, Grade 4: <25,000 cells/mm^3. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. An increase is defined as an increase in DAIDS grade relative to Baseline grade.
Time Frame: Baseline (Pre-dose, Day-1) and up to Day 35
Population: Safety Population. Only those participants with increase to grade 3 and increase to grade 4 were presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: GSK3640254 200 mg | Cohort 1: DRV/RTV 600/100 mg | Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg
Number analyzed (Participants) | 19 | 16 | 15
Participants
  Hemoglobin, Low, Increase to Grade 3 | 0 | 0 | 0
  Hemoglobin, Low, Increase to Grade 4 | 0 | 0 | 0
  Leukocytes, Low, Increase to Grade 3 | 0 | 0 | 0
  Leukocytes, Low, Increase to Grade 4 | 0 | 0 | 0
  Lymphocytes, Low, Increase to Grade 3 | 0 | 0 | 0
  Lymphocytes, Low, Increase to Grade 4 | 0 | 0 | 0
  Neutrophils, Low, Increase to Grade 3 | 0 | 0 | 0
  Neutrophils, Low, Increase to Grade 4 | 0 | 0 | 0
  Platelets, Low, Increase to Grade 3 | 0 | 0 | 0
  Platelets, Low, Increase to Grade 4 | 0 | 0 | 0

30. Secondary Outcome: Cohort 2: Number of Participants With Grade Increase Post-Baseline Relative to Baseline in Hematology Parameters
Description: Blood samples were collected for analysis of hematology parameters. Laboratory abnormalities were graded according to DAIDS grading table Version 2.1. For Hemoglobin Low, Grade 3: 7.0 to <9.0 g/dL (males) and 6.5 to <8.5 g/dL (females),Grade 4: <7.0 g/dL (males) and <6.5 g/dL (females); Leukocytes Low, Grade 3: 1000 to 1499 cells/mm^3,Grade 4: <1000 cells/mm^3; Lymphocytes Low, Grade 3: 350 to <500 cells/L,Grade 4: <350 cells/L; Neutrophils Low, Grade 3: 400 to 599 cells/mm^3, Grade 4: <400 cells/mm^3; Platelets Low, Grade 3: 25,000 to <50,000 cells/mm^3, Grade 4: <25,000 cells/mm^3. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. An increase is defined as an increase in DAIDS grade relative to Baseline grade.
Time Frame: Baseline (Pre-dose, Day-1) and up to Day 36
Population: Safety Population. Only those participants with increase to grade 3 and increase to grade 4 were presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: GSK3640254 200 mg | Cohort 2: ETR 200 mg | Cohort 2: GSK3640254 200 mg + ETR 200 mg
Number analyzed (Participants) | 19 | 16 | 16
Participants
  Hemoglobin, Low, Increase to Grade 3 | 0 | 0 | 0
  Hemoglobin, Low, Increase to Grade 4 | 0 | 0 | 0
  Leukocytes, Low, Increase to Grade 3 | 0 | 0 | 0
  Leukocytes, Low, Increase to Grade 4 | 0 | 0 | 0
  Lymphocytes, Low, Increase to Grade 3 | 0 | 0 | 0
  Lymphocytes, Low, Increase to Grade 4 | 0 | 0 | 0
  Neutrophils, Low, Increase to Grade 3 | 0 | 0 | 0
  Neutrophils, Low, Increase to Grade 4 | 0 | 0 | 0
  Platelets, Low, Increase to Grade 3 | 0 | 0 | 0
  Platelets, Low, Increase to Grade 4 | 0 | 0 | 0

31. Secondary Outcome: Cohort 3: Number of Participants With Grade Increase Post-Baseline Relative to Baseline in Hematology Parameters
Description: as for outcome 30
Time Frame: Baseline (Pre-dose, Day-1) and up to Day 26
Population: Safety Population. Only those participants with increase to grade 3 and increase to grade 4 were presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: GSK3640254 200 mg | Cohort 3: GSK3640254 200 mg+ DRV/RTV 600/100 mg+ ETR 200 mg
Number analyzed (Participants) | 16 | 15
Participants
  Hemoglobin, Low, Increase to Grade 3 | 0 | 0
  Hemoglobin, Low, Increase to Grade 4 | 0 | 0
  Leukocytes, Low, Increase to Grade 3 | 0 | 0
  Leukocytes, Low, Increase to Grade 4 | 0 | 0
  Lymphocytes, Low, Increase to Grade 3 | 0 | 0
  Lymphocytes, Low, Increase to Grade 4 | 0 | 0
  Neutrophils, Low, Increase to Grade 3 | 0 | 0
  Neutrophils, Low, Increase to Grade 4 | 0 | 0
  Platelets, Low, Increase to Grade 3 | 0 | 0
  Platelets, Low, Increase to Grade 4 | 0 | 0

32. Secondary Outcome: Cohort 1: Number of Participants With Grade Increase Post-Baseline Relative to Baseline in Clinical Chemistry Parameters: Alanine Aminotransferase, Albumin, Alkaline Phosphatase, Amylase, Aspartate Aminotransferase, Bilirubin and Direct Bilirubin
Description: Blood samples were collected for analysis of clinical chemistry parameters. Laboratory abnormalities were graded according to DAIDS grading table Version 2.1. For Alanine Aminotransferase High; Grade 3: 5.0 to <10.0 times (×) Upper Limit Normal (ULN), Grade 4: >=10.0 × ULN; Albumin Low, Grade 3: <2.0 grams per deciliter (g/dL), Grade 4: Not Applicable; Alkaline Phosphatase High, Grade 3: 5.0 to <10.0 × ULN, Grade 4: >=10.0 × ULN; Amylase High, Grade 3: 3.0 to <5.0 × ULN, Grade 4: >=5.0 × ULN; Aspartate Aminotransferase High, Grade 3: 5.0 to <10.0 × ULN, Grade 4: >=10.0 × ULN; Bilirubin High, Grade 3: 2.6 to<5.0 × ULN, Grade 4: >=5.0 × ULN and Direct Bilirubin High, Grade 3: >ULN with other signs and symptoms of hepatotoxicity, Grade 4: >ULN with life-threatening consequences. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. An increase is defined as an increase in DAIDS grade relative to Baseline grade.
Time Frame: Baseline (Pre-dose, Day-1) and up to Day 35
Population: Safety Population. Only those participants with increase to grade 3 and increase to grade 4 were presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: GSK3640254 200 mg | Cohort 1: DRV/RTV 600/100 mg | Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg
Number analyzed (Participants) | 19 | 16 | 15
Participants
  Alanine Aminotransferase, High, Increase to Grade 3 | 0 | 0 | 0
  Alanine Aminotransferase, High, Increase to Grade 4 | 0 | 0 | 0
  Albumin, Low, Increase to Grade 3 | 0 | 0 | 0
  Albumin, Low, Increase to Grade 4 | 0 | 0 | 0
  Alkaline Phosphatase, High, Increase to Grade 3 | 0 | 0 | 0
  Alkaline Phosphatase, High, Increase to Grade 4 | 0 | 0 | 0
  Amylase, High, Increase to Grade 3 | 0 | 0 | 0
  Amylase, High, Increase to Grade 4 | 0 | 0 | 0
  Aspartate Aminotransferase, High, Increase to Grade 3 | 0 | 0 | 0
  Aspartate Aminotransferase, High, Increase to Grade 4 | 0 | 0 | 0
  Bilirubin, High, Increase to Grade 3 | 0 | 0 | 0
  Bilirubin, High, Increase to Grade 4 | 0 | 0 | 0
  Direct Bilirubin, High, Increase to Grade 3 | 0 | 0 | 0
  Direct Bilirubin, High, Increase to Grade 4 | 0 | 0 | 0

33. Secondary Outcome: Cohort 1: Number of Participants With Grade Increase Post-Baseline Relative to Baseline in Clinical Chemistry Parameters: Calcium, Creatine Kinase, Creatinine, Phosphate, Potassium and Sodium
Description: Blood samples were collected for analysis of clinical chemistry parameters. Laboratory abnormalities were graded according to DAIDS grading table Version 2.1. For Calcium High, Grade 3: 12.5 to <13.5 milligrams/deciliter (mg/dL), Grade 4: >=13.5 mg/dL; Calcium Low, Grade 3: 6.1 to <7.0 mg/dL, Grade 4: <6.1 mg/dL; Creatine Kinase High, Grade 3: 10 to <20 × ULN, Grade 4: >=20 × ULN; Creatinine High, Grade 3: >1.8 to <3.5 ULN, Grade 4: >=3.5 × ULN; Phosphate Low, Grade 3: 1.0 to <1.4 mg/dL, Grade 4: <1.0 mg/dL; Potassium High, Grade 3: 6.5 to <7.0 Milliequivalents per liter (mEq/L),Grade 4: >=7.0 mEq/L; Potassium Low, Grade 3: 2.0 to <2.5 mEq/L, Grade 4: <2.00 mEq/L; Sodium High, Grade 3: 154 to <160 mEq/L, Grade 4:>=160 mEq/L; Sodium Low, Grade 3: 121 to <125 mEq/L, Grade 4:<=120 mEq/L. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. An increase is defined as an increase in DAIDS grade relative to Baseline grade.
Time Frame: Baseline (Pre-dose, Day-1) and up to Day 35
Population: Safety Population. Only those participants with increase to grade 3 and increase to grade 4 were presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: GSK3640254 200 mg | Cohort 1: DRV/RTV 600/100 mg | Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg
Number analyzed (Participants) | 19 | 16 | 15
Participants
  Calcium, Low, Increase to Grade 3 | 0 | 0 | 0
  Calcium, Low, Increase to Grade 4 | 0 | 0 | 0
  Calcium, High, Increase to Grade 3 | 0 | 0 | 0
  Calcium, High, Increase to Grade 4 | 0 | 0 | 0
  Creatine Kinase, High, Increase to Grade 3 | 0 | 0 | 0
  Creatine Kinase, High, Increase to Grade 4 | 0 | 0 | 0
  Creatinine, High, Increase to Grade 3 | 0 | 0 | 0
  Creatinine, High, Increase to Grade 4 | 0 | 0 | 0
  Phosphate, Low, Increase to Grade 3 | 0 | 0 | 0
  Phosphate, Low, Increase to Grade 4 | 0 | 0 | 0
  Potassium, Low, Increase to Grade 3 | 0 | 0 | 0
  Potassium, Low, Increase to Grade 4 | 0 | 0 | 0
  Potassium, High, Increase to Grade 3 | 0 | 0 | 0
  Potassium, High, Increase to Grade 4 | 0 | 0 | 0
  Sodium, Low, Increase to Grade 3 | 0 | 0 | 0
  Sodium, Low, Increase to Grade 4 | 0 | 0 | 0
  Sodium, High, Increase to Grade 3 | 0 | 0 | 0
  Sodium, High, Increase to Grade 4 | 0 | 0 | 0

34. Secondary Outcome: Cohort 1: Number of Participants With Grade Increase Post-Baseline Relative to Baseline in Clinical Chemistry Parameters: Glucose, Triglycerides, Lipase, Urate and Cholesterol
Description: Blood samples were collected for analysis of clinical chemistry parameters. Laboratory abnormalities were graded according to DAIDS grading table Version 2.1. For Glucose High, Grade 3: >250 to 500 mg/dL, Grade 4: >=500 mg/dL, Glucose Low, Grade 3: 30 to<40 mg/dL, Grade 4:<30 mg/dL; Triglycerides High, Grade 3: >500 to <1.000 mg/dL, Grade 4:>1000 mg/dL; Lipase High, Grade 3: 3.0 to <5.0×ULN, Grade 4:>=5.0×ULN; Urate High, Grade 3: 12.0 to <15.0 mEq/L, Grade 4:>=15.0 mEq/L; Cholesterol High, Grade 3: >=300 mg/dL, Grade 4: Not Applicable. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. An increase is defined as an increase in DAIDS grade relative to Baseline grade.
Time Frame: Baseline (Pre-dose, Day-1) and up to Day 35
Population: Safety Population. Only those participants with increase to grade 3 and increase to grade 4 were presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: GSK3640254 200 mg | Cohort 1: DRV/RTV 600/100 mg | Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg
Number analyzed (Participants) | 19 | 16 | 15
Participants
  Glucose, Low, Increase to Grade 3 | 0 | 0 | 0
  Glucose, Low, Increase to Grade 4 | 0 | 0 | 0
  Glucose, High, Increase to Grade 3 | 0 | 0 | 0
  Glucose, High, Increase to Grade 4 | 0 | 0 | 0
  Triglycerides, High, Increase to Grade 3 | 0 | 0 | 0
  Triglycerides, High, Increase to Grade 4 | 0 | 0 | 0
  Lipase, High, Increase to Grade 3 | 0 | 0 | 0
  Lipase, High, Increase to Grade 4 | 0 | 0 | 0
  Urate, High, Increase to Grade 3 | 0 | 0 | 0
  Urate, High, Increase to Grade 4 | 0 | 0 | 0
  Cholesterol, High, Increase to Grade 3 | 0 | 0 | 0
  Cholesterol, High, Increase to Grade 4 | 0 | 0 | 0

35. Secondary Outcome: Cohort 2: Number of Participants With Grade Increase Post-Baseline Relative to Baseline in Clinical Chemistry Parameters: Alanine Aminotransferase, Albumin, Alkaline Phosphatase, Amylase, Aspartate Aminotransferase, Bilirubin and Direct Bilirubin
Description: Blood samples were collected for analysis of clinical chemistry parameters. Laboratory abnormalities were graded according to DAIDS grading table Version 2.1. For Alanine Aminotransferase High; Grade 3: 5.0 to <10.0 × ULN, Grade 4: >=10.0 × ULN; Albumin Low, Grade 3: <2.0 g/dL, Grade 4: Not Applicable; Alkaline Phosphatase High, Grade 3: 5.0 to <10.0 × ULN, Grade 4: >=10.0 × ULN; Amylase High, Grade 3: 3.0 to <5.0 × ULN, Grade 4: >=5.0 × ULN; Aspartate Aminotransferase High, Grade 3: 5.0 to <10.0 × ULN, Grade 4: >=10.0 × ULN; Bilirubin High, Grade 3: 2.6 to<5.0 × ULN, Grade 4: >=5.0 × ULN and Direct Bilirubin High, Grade 3: >ULN with other signs and symptoms of hepatotoxicity, Grade 4: >ULN with life-threatening consequences. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. An increase is defined as an increase in DAIDS grade relative to Baseline grade.
Time Frame: Baseline (Pre-dose, Day-1) and up to Day 36
Population: Safety Population. Only those participants with increase to grade 3 and increase to grade 4 were presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: GSK3640254 200 mg | Cohort 2: ETR 200 mg | Cohort 2: GSK3640254 200 mg + ETR 200 mg
Number analyzed (Participants) | 19 | 16 | 16
Participants
  Alanine Aminotransferase, High, Increase to Grade 3 | 0 | 0 | 0
  Alanine Aminotransferase, High, Increase to Grade 4 | 0 | 0 | 0
  Albumin, Low, Increase to Grade 3 | 0 | 0 | 0
  Albumin, Low, Increase to Grade 4 | 0 | 0 | 0
  Alkaline Phosphatase, High, Increase to Grade 3 | 0 | 0 | 0
  Alkaline Phosphatase, High, Increase to Grade 4 | 0 | 0 | 0
  Amylase, High, Increase to Grade 3 | 0 | 0 | 0
  Amylase, High, Increase to Grade 4 | 0 | 0 | 0
  Aspartate Aminotransferase, High, Increase to Grade 3 | 0 | 0 | 0
  Aspartate Aminotransferase, High, Increase to Grade 4 | 0 | 0 | 0
  Bilirubin, High, Increase to Grade 3 | 0 | 0 | 0
  Bilirubin, High, Increase to Grade 4 | 0 | 0 | 0
  Direct Bilirubin, High, Increase to Grade 3 | 0 | 0 | 0
  Direct Bilirubin, High, Increase to Grade 4 | 0 | 0 | 0

36. Secondary Outcome: Cohort 2: Number of Participants With Grade Increase Post-Baseline Relative to Baseline in Clinical Chemistry Parameters: Calcium, Creatine Kinase, Creatinine, Phosphate, Potassium and Sodium
Description: Blood samples were collected for analysis of clinical chemistry parameters. Laboratory abnormalities were graded according to DAIDS grading table Version 2.1. For Calcium High, Grade 3: 12.5 to <13.5 mg/dL, Grade 4: >=13.5 mg/dL; Calcium Low, Grade 3: 6.1 to <7.0 mg/dL, Grade 4: <6.1 mg/dL; Creatine Kinase High, Grade 3: 10 to <20 × ULN, Grade 4: >=20 × ULN; Creatinine High, Grade 3: >1.8 to <3.5 ULN, Grade 4: >=3.5 × ULN; Phosphate Low, Grade 3: 1.0 to <1.4 mg/dL, Grade 4: <1.0 mg/dL; Potassium High, Grade 3: 6.5 to <7.0 mEq/L,Grade 4: >=7.0 mEq/L; Potassium Low, Grade 3: 2.0 to <2.5 mEq/L, Grade 4: <2.00 mEq/L; Sodium High, Grade 3: 154 to <160 mEq/L, Grade 4:>=160 mEq/L; Sodium Low, Grade 3: 121 to <125 mEq/L, Grade 4:<=120 mEq/L. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. An increase is defined as an increase in DAIDS grade relative to Baseline grade.
Time Frame: Baseline (Pre-dose, Day-1) and up to Day 36
Population: Safety Population. Only those participants with increase to grade 3 and increase to grade 4 presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: GSK3640254 200 mg | Cohort 2: ETR 200 mg | Cohort 2: GSK3640254 200 mg + ETR 200 mg
Number analyzed (Participants) | 19 | 16 | 16
Participants
  Calcium, Low, Increase to Grade 3 | 0 | 0 | 0
  Calcium, Low, Increase to Grade 4 | 0 | 0 | 0
  Calcium, High, Increase to Grade 3 | 0 | 0 | 0
  Calcium, High, Increase to Grade 4 | 0 | 0 | 0
  Creatine Kinase, High, Increase to Grade 3 | 0 | 0 | 0
  Creatine Kinase, High, Increase to Grade 4 | 0 | 0 | 0
  Creatinine, High, Increase to Grade 3 | 0 | 0 | 0
  Creatinine, High, Increase to Grade 4 | 0 | 0 | 0
  Phosphate, Low, Increase to Grade 3 | 0 | 0 | 0
  Phosphate, Low, Increase to Grade 4 | 0 | 0 | 0
  Potassium, Low, Increase to Grade 3 | 0 | 0 | 0
  Potassium, Low, Increase to Grade 4 | 0 | 0 | 0
  Potassium, High, Increase to Grade 3 | 0 | 0 | 0
  Potassium, High, Increase to Grade 4 | 0 | 0 | 0
  Sodium, Low, Increase to Grade 3 | 0 | 0 | 0
  Sodium, Low, Increase to Grade 4 | 0 | 0 | 0
  Sodium, High, Increase to Grade 3 | 0 | 0 | 0
  Sodium, High, Increase to Grade 4 | 0 | 0 | 0

37. Secondary Outcome: Cohort 2: Number of Participants With Grade Increase Post-Baseline Relative to Baseline in Clinical Chemistry Parameters: Glucose, Triglycerides, Lipase, Urate and Cholesterol
Description: as for outcome 34
Time Frame: Baseline (Pre-dose, Day-1) and up to Day 36
Population: Safety Population. Only those participants with increase to grade 3 and increase to grade 4 were presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: GSK3640254 200 mg | Cohort 2: ETR 200 mg | Cohort 2: GSK3640254 200 mg + ETR 200 mg
Number analyzed (Participants) | 19 | 16 | 16
Participants
  Glucose, Low, Increase to Grade 3 | 0 | 0 | 0
  Glucose, Low, Increase to Grade 4 | 0 | 0 | 0
  Glucose, High, Increase to Grade 3 | 0 | 0 | 0
  Glucose, High, Increase to Grade 4 | 0 | 0 | 0
  Triglycerides, High, Increase to Grade 3 | 0 | 0 | 0
  Triglycerides, High, Increase to Grade 4 | 0 | 0 | 0
  Lipase, High, Increase to Grade 3 | 0 | 0 | 0
  Lipase, High, Increase to Grade 4 | 0 | 0 | 0
  Urate, High, Increase to Grade 3 | 0 | 0 | 0
  Urate, High, Increase to Grade 4 | 0 | 0 | 0
  Cholesterol, High, Increase to Grade 3 | 0 | 0 | 0
  Cholesterol, High, Increase to Grade 4 | 0 | 0 | 0

38. Secondary Outcome: Cohort 3: Number of Participants With Grade Increase Post-Baseline Relative to Baseline in Clinical Chemistry Parameters: Alanine Aminotransferase, Albumin, Alkaline Phosphatase, Amylase, Aspartate Aminotransferase, Bilirubin and Direct Bilirubin
Description: as for outcome 35
Time Frame: Baseline (Pre-dose, Day-1) and up to Day 26
Population: Safety Population. Only those participants with increase to grade 3 and increase to grade 4 were presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: GSK3640254 200 mg | Cohort 3: GSK3640254 200 mg+ DRV/RTV 600/100 mg+ ETR 200 mg
Number analyzed (Participants) | 16 | 15
Participants
  Alanine Aminotransferase, High, Increase to Grade 3 | 0 | 0
  Alanine Aminotransferase, High, Increase to Grade 4 | 0 | 0
  Albumin, Low, Increase to Grade 3 | 0 | 0
  Albumin, Low, Increase to Grade 4 | 0 | 0
  Alkaline Phosphatase, High, Increase to Grade 3 | 0 | 0
  Alkaline Phosphatase, High, Increase to Grade 4 | 0 | 0
  Amylase, High, Increase to Grade 3 | 0 | 0
  Amylase, High, Increase to Grade 4 | 0 | 0
  Aspartate Aminotransferase, High, Increase to Grade 3 | 0 | 0
  Aspartate Aminotransferase, High, Increase to Grade 4 | 0 | 0
  Bilirubin, High, Increase to Grade 3 | 0 | 0
  Bilirubin, High, Increase to Grade 4 | 0 | 0
  Direct Bilirubin, High, Increase to Grade 3 | 0 | 0
  Direct Bilirubin, High, Increase to Grade 4 | 0 | 0

39. Secondary Outcome: Cohort 3: Number of Participants With Grade Increase Post-Baseline Relative to Baseline in Clinical Chemistry Parameters: Calcium, Creatine Kinase, Creatinine, Phosphate, Potassium and Sodium
Description: as for outcome 36
Time Frame: Baseline (Pre-dose, Day-1) and up to Day 26
Population: Safety Population. Only those participants with increase to grade 3 and increase to grade 4 were presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: GSK3640254 200 mg | Cohort 3: GSK3640254 200 mg+ DRV/RTV 600/100 mg+ ETR 200 mg
Number analyzed (Participants) | 16 | 15
Participants
  Calcium, Low, Increase to Grade 3 | 0 | 0
  Calcium, Low, Increase to Grade 4 | 0 | 0
  Calcium, High, Increase to Grade 3 | 0 | 0
  Calcium, High, Increase to Grade 4 | 0 | 0
  Creatine Kinase, High, Increase to Grade 3 | 0 | 0
  Creatine Kinase, High, Increase to Grade 4 | 0 | 0
  Creatinine, High, Increase to Grade 3 | 0 | 0
  Creatinine, High, Increase to Grade 4 | 0 | 0
  Phosphate, Low, Increase to Grade 3 | 0 | 0
  Phosphate, Low, Increase to Grade 4 | 0 | 0
  Potassium, Low, Increase to Grade 3 | 0 | 0
  Potassium, Low, Increase to Grade 4 | 0 | 0
  Potassium, High, Increase to Grade 3 | 0 | 0
  Potassium, High, Increase to Grade 4 | 0 | 0
  Sodium, Low, Increase to Grade 3 | 0 | 0
  Sodium, Low, Increase to Grade 4 | 0 | 0
  Sodium, High, Increase to Grade 3 | 0 | 0
  Sodium, High, Increase to Grade 4 | 0 | 0

40. Secondary Outcome: Cohort 3: Number of Participants With Grade Increase Post-Baseline Relative to Baseline in Clinical Chemistry Parameters: Glucose, Triglycerides, Lipase, Urate and Cholesterol
Description: as for outcome 34
Time Frame: Baseline (Pre-dose, Day-1) and up to Day 26
Population: Safety Population. Only those participants with increase to grade 3 and increase to grade 4 were presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: GSK3640254 200 mg | Cohort 3: GSK3640254 200 mg+ DRV/RTV 600/100 mg+ ETR 200 mg
Number analyzed (Participants) | 16 | 15
Participants
  Glucose, Low, Increase to Grade 3 | 0 | 0
  Glucose, Low, Increase to Grade 4 | 0 | 0
  Glucose, High, Increase to Grade 3 | 0 | 0
  Glucose, High, Increase to Grade 4 | 0 | 0
  Triglycerides, High, Increase to Grade 3 | 0 | 0
  Triglycerides, High, Increase to Grade 4 | 0 | 0
  Lipase, High, Increase to Grade 3 | 0 | 0
  Lipase, High, Increase to Grade 4 | 0 | 0
  Urate, High, Increase to Grade 3 | 0 | 0
  Urate, High, Increase to Grade 4 | 0 | 0
  Cholesterol, High, Increase to Grade 3 | 0 | 0
  Cholesterol, High, Increase to Grade 4 | 0 | 0

41. Secondary Outcome: Cohort 1: Number of Participants With Grade Increase Post-Baseline Relative to Baseline in Urinalysis Parameters
Description: Urine samples were collected for urinalysis parameters. Laboratory abnormalities were graded according to DAIDS grading table Version 2.1. For Erythrocytes High, Grade 3: Gross, with or without clots OR with Red Blood Cells (RBC) casts OR intervention indicated, Grade 4: Life-threatening consequences; Glucose High, Grade 3: >2+ (proportionate concentration by dipstick test) or >500 mg, Grade 4: >500 mg; Protein High, Grade 3: 3+ (proportionate concentration by dipstick test) or higher, Grade 4: Not Applicable. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. An increase is defined as an increase in DAIDS grade relative to Baseline grade.
Time Frame: Baseline (Pre-dose, Day-1) and up to Day 35
Population: Safety Population. Only those participants with increase to grade 3 and increase to grade 4 were presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: GSK3640254 200 mg | Cohort 1: DRV/RTV 600/100 mg | Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg
Number analyzed (Participants) | 19 | 16 | 15
Participants
  Erythrocytes, High, Increase to Grade 3 | 0 | 0 | 0
  Erythrocytes, High, Increase to Grade 4 | 0 | 0 | 0
  Glucose, High, Increase to Grade 3 | 0 | 0 | 0
  Glucose, High, Increase to Grade 4 | 0 | 0 | 0
  Protein, High, Increase to Grade 3 | 0 | 0 | 0
  Protein, High, Increase to Grade 4 | 0 | 0 | 0

42. Secondary Outcome: Cohort 2: Number of Participants With Grade Increase Post-Baseline Relative to Baseline in Urinalysis Parameters
Description: Urine samples were collected for urinalysis parameters. Laboratory abnormalities were graded according to DAIDS grading table Version 2.1. For Erythrocytes High, Grade 3: Gross, with or without clots OR with RBC casts OR intervention indicated, Grade 4: Life-threatening consequences; Glucose High, Grade 3: >2+ (proportionate concentration by dipstick test) or >500 mg, Grade 4: >500 mg; Protein High, Grade 3: 3+ (proportionate concentration by dipstick test) or higher, Grade 4: Not Applicable. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. An increase is defined as an increase in DAIDS grade relative to Baseline grade.
Time Frame: Baseline (Pre-dose, Day-1) and up to Day 36
Population: Safety Population. Only those participants with increase to grade 3 and increase to grade 4 were presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: GSK3640254 200 mg | Cohort 2: ETR 200 mg | Cohort 2: GSK3640254 200 mg + ETR 200 mg
Number analyzed (Participants) | 19 | 16 | 16
Participants
  Erythrocytes, High, Increase to Grade 3 | 0 | 0 | 0
  Erythrocytes, High, Increase to Grade 4 | 0 | 0 | 0
  Glucose, High, Increase to Grade 3 | 0 | 0 | 0
  Glucose, High, Increase to Grade 4 | 0 | 0 | 0
  Protein, High, Increase to Grade 3 | 0 | 0 | 0
  Protein, High, Increase to Grade 4 | 0 | 0 | 0

43. Secondary Outcome: Cohort 3: Number of Participants With Grade Increase Post-Baseline Relative to Baseline in Urinalysis Parameters
Description: as for outcome 42
Time Frame: Baseline (Pre-dose, Day-1) and up to Day 26
Population: Safety Population. Only those participants with increase to grade 3 and increase to grade 4 were presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: GSK3640254 200 mg | Cohort 3: GSK3640254 200 mg+ DRV/RTV 600/100 mg+ ETR 200 mg
Number analyzed (Participants) | 16 | 15
Participants
  Erythrocytes, High, Increase to Grade 3 | 0 | 0
  Erythrocytes, High, Increase to Grade 4 | 0 | 0
  Glucose, High, Increase to Grade 3 | 0 | 0
  Glucose, High, Increase to Grade 4 | 0 | 0
  Protein, High, Increase to Grade 3 | 0 | 0
  Protein, High, Increase to Grade 4 | 0 | 0

44. Secondary Outcome: Cohort 1: Number of Participants With Vital Sign Values of Potential Clinical Importance (PCI) Criteria
Description: Vital signs including systolic blood pressure (SBP), diastolic blood pressure (DBP) and pulse rate were measured in a supine position after atleast 5 minutes of rest. The PCI ranges for vitals were as follows; for SBP <85 or >140 millimeters of mercury (mmHg), for DBP <45 or >90 mmHg, for pulse rate <40 or >100 beats per minute. The number of participants with vital signs of PCI were presented.
Time Frame: Up to Day 35
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: GSK3640254 200 mg | Cohort 1: DRV/RTV 600/100 mg | Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg
Number analyzed (Participants) | 19 | 16 | 15
Participants
  SBP | 0 | 2 | 0
  DBP | 0 | 0 | 0
  Pulse rate | 0 | 0 | 0

45. Secondary Outcome: Cohort 2: Number of Participants With Vital Sign Values of PCI Criteria
Description: Vital signs including SBP, DBP and pulse rate were measured in a supine position after atleast 5 minutes of rest. The PCI ranges for vitals were as follows; for SBP <85 or >140 mmHg, for DBP <45 or >90 mmHg, for pulse rate <40 or >100 beats per minute. The number of participants with vital signs of PCI were presented.
Time Frame: Up to Day 36
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: GSK3640254 200 mg | Cohort 2: ETR 200 mg | Cohort 2: GSK3640254 200 mg + ETR 200 mg
Number analyzed (Participants) | 19 | 16 | 16
Participants
  SBP | 0 | 0 | 0
  DBP | 0 | 0 | 1
  Pulse rate | 0 | 0 | 0

46. Secondary Outcome: Cohort 3: Number of Participants With Vital Sign Values of PCI Criteria
Description: as for outcome 45
Time Frame: Up to Day 26
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: GSK3640254 200 mg | Cohort 3: GSK3640254 200 mg+ DRV/RTV 600/100 mg+ ETR 200 mg
Number analyzed (Participants) | 16 | 15
Participants
  SBP | 1 | 0
  DBP | 0 | 0
  Pulse rate | 0 | 0

47. Secondary Outcome: Cohort 1: Number of Participants With Clinically Significant Abnormal Electrocardiogram (ECG) Findings
Description: A 12-lead ECG was recorded with the participant in a supine position using an automated ECG machine. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for number of participants with clinically significant abnormal ECG findings were reported. Data has been presented for the participants with respect to the actual treatment received in respective treatment periods.
Time Frame: Day 1 (2,4,6 Hours), Day 7 and Day 11 in Treatment Period 1; Day 12 (2,4,6 Hours), Day 21 in Treatment Period 2; Day 22 (2,4,6 Hours), Day 26 and Day 35 in Treatment Period 3
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: GSK3640254 200 mg | Cohort 1: DRV/RTV 600/100 mg | Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg
Number analyzed (Participants) | 19 | 16 | 15
Participants
  2 Hours, Day 1: number analyzed (Participants) | 19 | 0 | 0
  2 Hours, Day 1 | 0 |  |
  4 Hours, Day 1: number analyzed (Participants) | 19 | 0 | 0
  4 Hours, Day 1 | 0 |  |
  6 Hours; Day 1: number analyzed (Participants) | 19 | 0 | 0
  6 Hours; Day 1 | 0 |  |
  Day 7: number analyzed (Participants) | 19 | 0 | 0
  Day 7 | 0 |  |
  Day 11: number analyzed (Participants) | 16 | 0 | 0
  Day 11 | 0 |  |
  2 Hours, Day 12: number analyzed (Participants) | 0 | 16 | 0
  2 Hours, Day 12 |  | 0 |
  4 Hours, Day 12: number analyzed (Participants) | 0 | 16 | 0
  4 Hours, Day 12 |  | 0 |
  6 Hours; Day 12: number analyzed (Participants) | 0 | 16 | 0
  6 Hours; Day 12 |  | 0 |
  Day 21: number analyzed (Participants) | 0 | 16 | 0
  Day 21 |  | 0 |
  2 Hours; Day 22: number analyzed (Participants) | 0 | 0 | 15
  2 Hours; Day 22 |  |  | 0
  4 Hours; Day 22: number analyzed (Participants) | 0 | 0 | 15
  4 Hours; Day 22 |  |  | 0
  6 Hours; Day 22: number analyzed (Participants) | 0 | 0 | 15
  6 Hours; Day 22 |  |  | 0
  Day 26: number analyzed (Participants) | 0 | 0 | 15
  Day 26 |  |  | 0
  Day 35: number analyzed (Participants) | 0 | 0 | 15
  Day 35 |  |  | 0

48. Secondary Outcome: Cohort 2: Number of Participants With Clinically Significant Abnormal ECG Findings
Description: as for outcome 47
Time Frame: Day 1 (2,4,6 Hours), Day 7 and Day 11 in Treatment Period 1; Day 12 (2,4,6 Hours), Day 21 in Treatment Period 2; Day 22 (2,4,6 Hours), Day 26 and Day 36 in Treatment Period 3
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: GSK3640254 200 mg | Cohort 2: ETR 200 mg | Cohort 2: GSK3640254 200 mg + ETR 200 mg
Number analyzed (Participants) | 19 | 16 | 16
Participants
  2 Hours, Day 1: number analyzed (Participants) | 19 | 0 | 0
  2 Hours, Day 1 | 0 |  |
  4 Hours, Day 1: number analyzed (Participants) | 19 | 0 | 0
  4 Hours, Day 1 | 0 |  |
  6 Hours; Day 1: number analyzed (Participants) | 19 | 0 | 0
  6 Hours; Day 1 | 0 |  |
  Day 7: number analyzed (Participants) | 19 | 0 | 0
  Day 7 | 0 |  |
  Day 11: number analyzed (Participants) | 16 | 0 | 0
  Day 11 | 0 |  |
  2 Hours, Day 12: number analyzed (Participants) | 0 | 16 | 0
  2 Hours, Day 12 |  | 0 |
  4 Hours, Day 12: number analyzed (Participants) | 0 | 16 | 0
  4 Hours, Day 12 |  | 0 |
  6 Hours; Day 12: number analyzed (Participants) | 0 | 16 | 0
  6 Hours; Day 12 |  | 0 |
  Day 21: number analyzed (Participants) | 0 | 16 | 0
  Day 21 |  | 0 |
  2 Hours; Day 22: number analyzed (Participants) | 0 | 0 | 16
  2 Hours; Day 22 |  |  | 0
  4 Hours; Day 22: number analyzed (Participants) | 0 | 0 | 16
  4 Hours; Day 22 |  |  | 0
  6 Hours; Day 22: number analyzed (Participants) | 0 | 0 | 16
  6 Hours; Day 22 |  |  | 0
  Day 26: number analyzed (Participants) | 0 | 0 | 16
  Day 26 |  |  | 0
  Day 36: number analyzed (Participants) | 0 | 0 | 14
  Day 36 |  |  | 0

49. Secondary Outcome: Cohort 3: Number of Participants With Clinically Significant Abnormal ECG Findings
Description: as for outcome 47
Time Frame: Day 1 (2,4,6 Hours) in Treatment Period 1; Day 8 (2,4,6 Hours), Day 9 (2,4,6 Hours), Day 26 in Treatment Period 2
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: GSK3640254 200 mg | Cohort 3: GSK3640254 200 mg+ DRV/RTV 600/100 mg+ ETR 200 mg
Number analyzed (Participants) | 16 | 15
Participants
  2 Hours, Day 1: number analyzed (Participants) | 16 | 0
  2 Hours, Day 1 | 0 |
  4 Hours, Day 1: number analyzed (Participants) | 16 | 0
  4 Hours, Day 1 | 0 |
  6 Hours, Day 1: number analyzed (Participants) | 16 | 0
  6 Hours, Day 1 | 0 |
  2 Hours, Day 8: number analyzed (Participants) | 0 | 15
  2 Hours, Day 8 |  | 0
  4 Hours, Day 8: number analyzed (Participants) | 0 | 15
  4 Hours, Day 8 |  | 0
  6 Hours, Day 8: number analyzed (Participants) | 0 | 15
  6 Hours, Day 8 |  | 0
  2 Hours; Day 9: number analyzed (Participants) | 0 | 15
  2 Hours; Day 9 |  | 0
  4 Hours; Day 9: number analyzed (Participants) | 0 | 15
  4 Hours; Day 9 |  | 0
  6 Hours; Day 9: number analyzed (Participants) | 0 | 15
  6 Hours; Day 9 |  | 0
  Day 26: number analyzed (Participants) | 0 | 14
  Day 26 |  | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events (SAE) and non-serious adverse events (non-SAE) were collected up to Day 35 during Cohort 1; up to Day 36 during Cohort 2; up to Day 26 during Cohort 3
Description: Safety Population was used to assess all-cause mortality, SAE and non-SAE which comprised of all participants who received at least 1 dose of study medication. AEs were presented cohort-wise and treatment-wise.
Arm/Group | Cohort 1: GSK3640254 200 mg | Cohort 1: DRV/RTV 600/100 mg | Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg | Cohort 2: GSK3640254 200 mg | Cohort 2: ETR 200 mg | Cohort 2: GSK3640254 200 mg + ETR 200 mg | Cohort 3: GSK3640254 200 mg | Cohort 3: GSK3640254 200 mg+ DRV/RTV 600/100 mg+ ETR 200 mg
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/16 | 0/15 | 0/19 | 0/16 | 0/16 | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/16 | 0/15 | 0/19 | 0/16 | 0/16 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 6/19 | 4/16 | 5/15 | 3/19 | 4/16 | 7/16 | 1/16 | 8/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: GSK3640254 200 mg (N=19) | Cohort 1: DRV/RTV 600/100 mg (N=16) | Cohort 1: GSK3640254 200 mg + DRV/RTV 600/100 mg (N=15) | Cohort 2: GSK3640254 200 mg (N=19) | Cohort 2: ETR 200 mg (N=16) | Cohort 2: GSK3640254 200 mg + ETR 200 mg (N=16) | Cohort 3: GSK3640254 200 mg (N=16) | Cohort 3: GSK3640254 200 mg+ DRV/RTV 600/100 mg+ ETR 200 mg (N=15)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (3)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Scleral hyperaemia (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Application site irritation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT04630002/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/02/NCT04630002/SAP_001.pdf